CLINICAL TRIAL: NCT07258511
Title: A Phase 3 Randomized Study Comparing JNJ-79635322 and an Anti-BCMAxCD3 Bispecific Antibody in Participants With Relapsed or Refractory Multiple Myeloma Who Have Received at Least 3 Prior Lines of Therapy Including a PI, an IMiD, and an Anti CD38 Antibody
Brief Title: A Study Comparing JNJ-79635322 and an Anti-B-cell Maturation Antigen (BCMA)xCD3 Bispecific Antibody in Participants With Relapsed or Refractory Multiple Myeloma
Acronym: TRIlogy-4
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 79635322MMY3001; 79635322MMY3001 (Other: Janssen Research & Development, LLC); 2025-522007-18-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JNJ-79635322 (Experimental): Participants will receive subcutaneous (SC) dose of JNJ-79635322 until progressive disease (PD) or intolerable toxicity.
  Interventions: Drug: JNJ-79635322
- Anti BCMAxCD3 Bispecific Antibody (Active Comparator): Participants will receive teclistamab (an Anti BCMAxCD3 bispecific anitbody) as a SC injection until PD or intolerable toxicity.
  Interventions: Drug: Teclistamab

INTERVENTIONS:
Drug: JNJ-79635322 — JNJ-79635322 will be administered as SC injection.
  Arms: JNJ-79635322
Drug: Teclistamab — Teclistamab will be administered as SC injection.
  Arms: Anti BCMAxCD3 Bispecific Antibody

SUMMARY:
The purpose of this study is to evaluate how well JNJ-79635322 works when compared with an anti-B-cell maturation antigen (BCMA)xCD3 bispecific antibody.

ELIGIBILITY:
Inclusion:

* Documented diagnosis of multiple myeloma (MM) as defined by the criteria below:

  1. MM diagnosis according to the international myeloma working group (IMWG) diagnostic criteria
  2. Measurable disease at screening as assessed by central laboratory
* Received at least 3 prior lines of antimyeloma therapy including a proteasome inhibitor (PI), an immunomodulatory drug (IMiD), and an anti-cluster of differentiation (CD)38 antibody
* Documented evidence of progressive disease (PD) or failure to achieve a response (that is partial response [PR] or better) to the last line of therapy based on investigator's determination of response by IMWG criteria
* Have discontinued concurrent use of any other anticancer treatment (including nonpalliative radiotherapy) or investigational agent
* Have an eastern cooperative oncology group (ECOG) performance status of 0 to 2 at screening and immediately before the start of study treatment administration

Exclusion:

* Active hepatitis of infectious origin
* Known active or prior central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of MM
* Suspected or known allergies, hypersensitivity, or intolerance to the excipients of JNJ-79635322 and Teclistamab
* Major surgery , (example, requiring general anesthesia) within 2 weeks before first dose, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study
* Received or plans to receive any live, attenuated vaccine within 4 weeks before the first dose of study treatment, during, or within 90 days after the last dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-02-04 (Actual); Primary Completion 2028-12-12 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 5 years and 4 months
  ORR is defined as the percentage of participants who achieve partial response (PR) or better, according to the international myeloma working group (IMWG) response criteria.
Progression-Free Survival (PFS) | Up to 5 years and 4 months
  PFS is defined as the duration from the date of randomization to either progressive disease (PD) or death, whichever comes first. Disease progression will be determined according to the IMWG response criteria.

SECONDARY OUTCOMES:
Very Good Partial Response (VGPR) or Better | Up to 5 years and 4 months
  VGPR or better is defined as the percentage of participants achieving VGPR, complete response (CR), or stringent complete response (sCR) prior to subsequent antimyeloma therapy in accordance with the IMWG criteria during or after the study treatment.
Complete Response (CR) or Better | Up to 5 years and 4 months
  CR or better is defined as the percentage of participants achieving CR or sCR prior to subsequent antimyeloma therapy in accordance with the IMWG criteria during or after the study treatment.
Duration of Response (DoR) | Up to 5 years and 4 months
  DoR is defined as the time interval between the date of initial documentation of a response (partial response [PR] or better) to the date of first documented evidence of progressive disease according to the IMWG response criteria or death due to any cause, whichever occurs first.
Minimal Residual Disease (MRD)-negative CR | Up to 5 years and 4 months
  MRD-negative CR is defined as the percentage of participants who achieve MRD-negative status, as determined by next-generation flow cytometry (NGF), at any time point after randomization and prior to PD or subsequent antimyeloma therapy and who achieve CR or better.
MRD-negative CR at 9 months | 9 months
  MRD-negative CR at 9 months is defined as the participants who achieve MRD-negative status at 9 months, as determined by NGF prior to PD or subsequent anti-myeloma therapy and who also achieve CR or better, according to IMWG criteria.
Sustained MRD-negative CR | Up to 5 years and 4 months
  Sustained MRD-negative CR is defined as participants with confirmed CR or better who sustain MRD-negative status, as determined by NGF, for at least 12 months without any examination showing MRD-positive status or progressive disease in between.
Progression-Free Survival on the First Subsequent Line of Antimyeloma Therapy (PFS2) | Up to 5 years and 4 months
  PFS2 is defined as the time interval between the date of randomization and date of event, which is defined as progressive disease as assessed by investigator on the first subsequent line of antimyeloma therapy, or death from any cause, whichever occurs first. Those who are alive and for whom a second disease progression has not been observed are censored at the last date of follow-up.
Overall Survival (OS) | Up to 5 years and 4 months
  OS is defined as the time from the date of randomization to the date of the participant's death due to any cause.
Time To Next Line of Therapy (TTNT) | Up to 5 years and 4 months
  TTNT is defined as the time from randomization to the start of subsequent antimyeloma treatment. Death due to progressive disease without the start of any subsequent antimyeloma therapy will be considered as an event.
Number of Participants With Treatment-Emergent Adverse Events (TEAE) by Severity | Up to 5 years and 4 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment. Any new or worsening AE occurring at or after the initial administration of study treatment through the day of last dose plus 30 days or prior to the start of subsequent anticancer therapy, whichever is earlier, or any follow-up AE with onset date and time beyond 30 days after the last dose of study treatment but prior to the start of subsequent therapy or any AE that is considered treatment-related regardless of the start date of the event is considered to be treatment-emergent. TEAEs will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 6.0. Severity scale ranges from Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening, to Grade 5= death related to adverse event.
Number of Participants with Abnormalities in Clinical Laboratories Results | Up to 5 years and 4 months
  Number of participants with abnormalities in clinical laboratories results (serum chemistry and hematology) will be reported.
Change from Baseline in Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by Multiple Myeloma Symptom and Impact Questionnaire (MySIm-Q) Score | Baseline up to 5 years and 4 months
  Change from baseline in symptoms, functioning, and health-related quality of life (HRQoL) as assessed by multiple myeloma symptom and impact questionnaire (MySIm-Q) score will be reported. The MySIm-Q is a disease-specific patient-reported outcome (PRO) assessment with established content validity for participants with relapsed or refractory multiple myeloma (RRMM) and newly diagnosed MM.
Change from Baseline in Symptoms, Functioning, and HRQoL as Assessed by European Organization for Research and Treatment of Cancer Quality of life Questionnaire Core 30 (EORTC-QLQ-C30) Score | Baseline up to 5 years and 4 months
  Change from baseline in symptoms, functioning, and HRQoL as assessed by european organization for research and treatment of cancer quality of life questionnaire core 30 (EORTC-QLQ-C30) score will be reported.
Change from Baseline in Symptoms, Functioning, and HRQoL as Assessed by European Quality of Life 5-Dimensions 5-Level Version (EQ-5D-5L) Score | Baseline up to 5 years and 4 months
  The EQ-5D-5L is a generic measure of health status that contains 5-item questionnaire that assesses 5 domains (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). The scores for the 5 dimensions are used to compute a single utility score, ranging from zero (0.0) to 1 (1.0), representing the general health status of the individual.
Time to Worsening in Symptoms, Functioning, and HRQoL as Assessed by MySIm-Q Score | Up to 5 years and 4 months
  Time to worsening in symptoms, functioning, and HRQoL as assessed by MySIm-Q score will be reported. The MySIm-Q is a disease-specific PRO assessment with established content validity for participants with RRMM and newly diagnosed MM.
Time to Worsening in Symptoms, Functioning, and HRQoL as Assessed by EORTC-QLQ-C30 Score | Up to 5 years and 4 months
  Time to worsening in symptoms, functioning, and HRQoL as assessed by EORTC-QLQ-C30 score will be reported.
Time to Worsening in Symptoms, Functioning, and HRQoL as Assessed by EQ-5D-5L Score | Up to 5 years and 4 months
  The EQ-5D-5L is a generic measure of health status that contains 5-item questionnaire that assesses 5 domains (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). The scores for the 5 dimensions are used to compute a single utility score, ranging from zero (0.0) to 1 (1.0), representing the general health status of the individual.
Percentage of Participants With Meaningful Improvement in Symptoms, Functioning, and HRQoL as Assessed by MySIm-Q Score | Up to 5 years and 4 months
  The MySIm-Q is a disease-specific PRO assessment with established content validity for participants with RRMM and newly diagnosed MM. It is included to be complementary to the EORTC-QLQ-C30. It includes 17 items resulting in a symptom subscale and an impact subscale. The recall period is the "past 7 days" and responses are reported on a 5-point verbal rating scale.
Percentage of Participants With Meaningful Improvement in Symptoms, Functioning, and HRQoL as Assessed by EORTC-QLQ-C30 Score | Up to 5 years and 4 months
  Percentage of participants with meaningful improvement in symptoms, functioning, and HRQoL as assessed by EORTC-QLQ-C30 score will be reported.
Percentage of Participants With Meaningful Improvement in Symptoms, Functioning, and HRQoL as Assessed by EQ-5D-5L Score | Up to 5 years and 4 months
  The EQ-5D-5L is a generic measure of health status that contains 5-item questionnaire that assesses 5 domains (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). The scores for the 5 dimensions are used to compute a single utility score, ranging from zero (0.0) to 1 (1.0), representing the general health status of the individual.
Percentage of Participants With Side Effects Burden on the European Organization for Research and Treatment of Cancer Item List 46 (EORTC IL46) | Up to 5 years and 4 months
  Percentage of participants with side effects burden on the EORTC IL46 will be reported. The EORTC IL46 measures the global impression of burden due to treatment-related symptoms.
Serum Concentrations for JNJ-79635322 | Up to 5 years and 4 months
  Serum concentrations of JNJ-79635322 will be reported.
Number of Participants With Anti-drug Antibodies (ADA) to JNJ-79635322 | Up to 5 years and 4 months
  Serum samples will be analyzed for the detection of ADA to JNJ-79635322 using a validated assay method.
Number of Participants With Neutralizing Antibodies (NAb) to JNJ-79635322 | Up to 5 years and 4 months
  Number of participants who are ADA-positive will be assessed for the presence of NAbs.

CONTACTS AND LOCATIONS:
Locations (9):
- Australia (3):
  - Box Hill Hospital, Box Hill
  - Mater Hospital Brisbane, South Brisbane
  - Gold Coast University Hospital, Southport
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek MC, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Baruch Padeh MC, Ramat Poriya

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency